CLINICAL TRIAL: NCT01732081
Title: Hepatitis B Cohort: Predictive Factors of the Outcome of Chronic Hepatitis B Virus Infection
Brief Title: "Real-life" Cohort of Patients With Chronic Hepatitis B Virus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5452
Record Dates: First submitted 2012-11-16; First posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with chronic hepatitis B virus infection: Patients chronically infected with hepatitis B virus (HBV), and followed in university hospital of Strasbourg, France

SUMMARY:
It is estimated that 350-400 million people worldwide are chronically infected with hepatitis B virus (HBV). Cirrhosis and hepatocellular carcinoma are major complications of chronic HBV infection and are responsible of about 500,000 deaths each year. Although some predictive factors of the outcome of chronic HBV infection were reported, it remains needed to more precisely determine the factors which are associated with the outcome in non-selected patients. Indeed, these factors should help to identify patients who are likely to have a better or worse evolution of their chronic HBV infection over time and thus, to adapt their clinical management and monitoring.Therefore, our purpose is to constitute a "real-life" cohort of non-selected patients to create a database of epidemiological, clinical, biological, virological and therapeutic parameters, in order to determine factors associated with the outcome of chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic HBV infection (defined as HBsAg positive for at least 6 months)

Exclusion Criteria:

* Co-infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) and/or hepatitis D virus (HDV)
* Decompensated cirrhosis
* History of liver transplantation
* History of hepatocellular carcinoma (HCC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients chronically infected with hepatitis B virus (HBV), and followed in university hospital of Strasbourg, France
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
to determine factors associated with the outcome of chronic HBV infection | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France